CLINICAL TRIAL: NCT05971758
Title: Fimepinostat, Combination HDAC and Pi3-kinase Inhibitor Tumor-Directed Therapy for Cushing Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Anthony P. Heaney, Professor-in-Residence, Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FD-07548-01-A1; R01FD007548-01A1 (FDA)
Record Dates: First submitted 2023-07-06; First posted 2023-08-02 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Cushing Disease
MeSH Terms: conditions — Pituitary ACTH Hypersecretion | interventions — fimepinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fimepinostat 60mg (Active Comparator): two 30mg capsules once a day, 10 subjects
  Interventions: Drug: Fimepinostat
- Fimepinostat 30mg (Active Comparator): single 30mg capsule daily in 10 subjects
  Interventions: Drug: Fimepinostat

INTERVENTIONS:
Drug: Fimepinostat — The study will allow us to determine the efficacy and safety of these doses in the treatment of Cushing Disease (CD) and guide dose selection for subsequent, larger studies.

SUMMARY:
Supported by the pre-clinical data (summarized in Research Strategy), the investigators propose that Fimepinostat is an ideal candidate drug in the treatment and intervention of patients with Cushing Disease. The investigators propose a pilot, short-term (4 weeks) phase II single-center study to demonstrate the safety and efficacy of Fimepinostat in the treatment of patients with de novo, persistent, and/or recurrent CD recruited at the University of California, Los Angeles. The trial will have a 2-arm design and will simultaneously examine two different doses of Fimepinostat. The study will allow the investigators to determine the efficacy and safety of these doses in the treatment of CD and guide dose selection for subsequent, larger studies. Funding Source - FDA OOPD.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients at least 18 years old
* Patients with confirmed pituitary origin Cushing syndrome defined as 1, 2& 3 or 4 & 5 below:

  1. Persistent hypercortisolism defined as a mean of 3 consecutive 24h UFC at baseline assessment ≥ 1.3x ULN
  2. Normal or elevated plasma ACTH levels
  3. Pituitary adenoma > 4mm visible on MRI or inferior petrosal sinus sampling (IPSS) central to peripheral ACTH gradient >2 at baseline and/or >2 after DDAVP stimulation.
  4. Recurrent or persistent CD defined as pathologically confirmed previously resected pituitary ACTH-secreting tumor, and 24 hour UFC >ULN at least 4 weeks after pituitary surgery.
  5. Patients on medical treatment for CD. Washout periods will be completed as below before screening: Inhibitors of steroidogenesis (metyrapone, ketoconazole, osilodristat,

     * Levo-ketoconazole): 2 weeks
     * SRLs (pasireotide): 2 weeks
     * Progesterone receptor antagonist (mifepristone): 2 weeks
     * Dopamine agonists (cabergoline): 4 weeks
     * CYP3A4 strong inducers or inhibitors: varies between drugs; minimum 5-6 times the half-life of drug

Exclusion Criteria:

* Patients with compromised visual fields, or evidence of visual changes within past 6 months
* Patients with sellar tumor abutting or compressing the optic chiasm on MRI and normal visual fields
* Patients with Cushing's syndrome not due to an ACTH-secreting pituitary tumor
* Patients who have undergone major surgery including pituitary surgery within 1 month of screening or who have any major surgical procedures planned across the study period
* Patients with serum potassium < 3.5 mEq/L unless stably controlled on potassium supplementation
* Patients with poorly-controlled Diabetes mellitus evidenced by HbA1c levels >8
* Patients with poorly controlled hypertension (i.e. blood pressure ≥ 160/100 mm Hg)
* Patients who have clinically significant cardiovascular impairment, as evidenced by the presence of bradycardia, ventricular tachycardia, history of myocardial infarction within past year, or any other cardiovascular impairment that may pose significant health risk in view of the investigator.
* Patients with liver disease or history of liver disease such as cirrhosis, chronic active hepatitis B and C, or chronic persistent hepatitis, or patients with ALT or AST >1.5 x ULN, serum total bilirubin >ULN, serum albumin <0.67 x LLN at screening
* Patients with renal disease or history of renal disease with creatinine clearance of 30 cm3/min or less and/or creatinine > 1.5 mg/dl at screening
* Patients not biochemically euthyroid. Patients receiving thyroid-replacement therapy must be on a stable dose for at least 3 months.
* Patients who are known to be positive for HIV, or any other condition that significantly compromises subject's immune system.
* History of alcohol abuse or illicit substance use within past year.
* Female patients who are pregnant or lactating or are of childbearing potential unless willing to practice acceptable method of birth control. Women participating in the trial must employ double barrier method through oral contraceptive or diaphragm with partner utilizing a condom. Abstinence is an acceptable form of birth control if routinely practiced. Male participants must utilize a condom with spermicidal cap/jelly and agree to not donate sperm for up to 3 months beyond main study period.
* Patients who have participated in any clinical investigation with an investigational drug within 1 month prior to screening or within 5 half-lives of the investigational treatment whichever is longer.
* Patients with concomitant treatment of strong CYP3A4 inducers or inhibitors.
* Patients who have received pituitary irradiation within the last 5 years prior to the baseline visit
* Patients with known hepatitis B surface antigen (HbsAg) positivity
* Patients with known hepatitis C antibody (anti-HCV) positivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with mUFC ≤ 1.0xULN | Baseline, 4 weeks
  4 week UFC calculated as the mean of three 24h UFC specimens collected on consecutive days between day 24-28

SECONDARY OUTCOMES:
Number of participants with normalization (values within normal limits) or >50% improvement from baseline in 24h UFC, plasma ACTH, serum and salivary cortisol levels | Baseline, 4 weeks
  4 week UFC calculated as the mean of three 24h UFC specimens collected on consecutive days between day 24-28
body weight change from baseline | Baseline, Day 28
body mass index change from baseline | Baseline, Day 28
Systolic and Diastolic Blood Pressure Change from baseline | Baseline, Day 28
Cushing Disease health-related quality of life questionnaire (CushingQoL) change from baseline | Baseline, Day 28
  The CushingQoL is scored using a total score ranging from 0 to 100 with lower scores indicating a greater impact on QoL
Beck Depression inventory second edition (BDIII) change from baseline | Baseline, Day 28
  Beck Depression scale is scored as follows 1-10 These ups and downs are considered normal. 11-16 Mild mood disturbances. 17-20 borderline clinical depression. 21-30 Moderate depression. 31-40 Severe depression

CONTACTS AND LOCATIONS:
Locations (1):
- Ronald Reagan Medical Center, Los Angeles, California, United States